CLINICAL TRIAL: NCT03769272
Title: Optimal Left Ventricular Lead Positioning During Cardiac Resynchronisation Therapy; Comparison of Two Methods of Targeting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peter J Pugh (Other)
Responsible Party: Sponsor-Investigator, Peter J Pugh, Consultant Cardiologist, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 227862
Record Dates: First submitted 2018-08-19; First posted 2018-12-07 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Echocardiographic targeting
- Electrogram targeting
  Interventions: Procedure: Measurement of electrical delay during LV lead placement

INTERVENTIONS:
Procedure: Measurement of electrical delay during LV lead placement — Measurement of electrical signal in the heart during implantation of CRT, by positioning the lead in different places in the heart.
  Groups: Electrogram targeting

SUMMARY:
Cardiac Resynchronisation Therapy (CRT) is a well-known treatment for patients with heart failure. It is a special pacemaker that consists of three pacing wires, which are implanted in the right upper and bottom chambers of the heart and via a vein on the surface of the main pumping chamber (left bottom chamber). CRT helps by improving co- ordination between the top and the bottom chambers of the heart. By stimulating the heart from the left and right bottom chambers, co-ordination can be restored and heart function as well as symptoms improve. It is known that up to 30-40% of patients of patients undergoing CRT pacemaker implantation do not attain any benefit. Given the inherent risks and costs of pacemaker implantation and maintenance, a reduction in the rate of CRT "non-responders" is an important goal.

It has been suggested that presence of scar tissue in the heart and suboptimal placement of the pacing wire on the top of the main pumping chamber can explain this poor response. The best place to position the pacing wire on the surface of the main pumping chamber is the area that contracts last and it can be identified using ultrasound scan of the heart.

Unfortunately, ultrasound is not always possible to help identifying the best area and only a minority of hospitals are able to use this method. Therefore we aim to investigate alternative ways of positioning the pacing wire in the best possible area of the main pumping heart chamber. Investigators propose to measure electrical signals as an alternative and more effective way in positioning the wire in the most effective area. Investigators aim to look at the relationship between the best area identified by ultrasound scan and by electrical signals and also use electrical signals to avoid areas of scar.

DETAILED DESCRIPTION:
Cardiac Resynchronisation Therapy (CRT) reduces both morbidity and mortality in selected patients with left ventricular dysfunction and intraventricular conduction delay who remain symptomatic despite optimal medical therapy.

It is known that up to 30% of patients of patients undergoing CRT implantation do not attain symptomatic benefit . Given the inherent risks and costs of device implantation and maintenance, a reduction in the rate of CRT "non-responders" is an important goal.

Factors associated with a poor outcome include presence of myocardial scar, and suboptimal Left Ventricular (LV) lead placement.

Pacing the LV at the most delayed LV region promotes contractile synchrony resulting in more effective and energetically efficient ejection, geometric remodelling with reduced LV end-systolic volume and improved cardiac function.

Studies using transthoracic echocardiographic (TTE) parameters to target the LV lead positioning have shown that an optimal LV lead position at the site of latest mechanical activation, avoiding low strain amplitude (scar), was associated with superior response to CRT and improved survival that persisted during follow-up.

It remains unclear whether the site of latest mechanical activation is related to the site of latest electrical activation, nor whether sensed electrical signals correspond to sites of scar. The site of latest electrical activation is assessed during CRT implant by measuring electrical activation (LV electrical delay) of the LV at different sites in relation to the first deflection of the QRS complex of the surface electrocardiogram (ECG).

A recent study evaluated the relationship between LV electrical delay and CRT outcomes/ response to CRT and concluded that electrical dyssynchrony was strongly and independently associated with reverse remodelling and led to improvement in the Quality of Life with CRT.

Despite TTE being an effective way of assessing optimal LV lead positioning for identifying mechanical activation, it is expensive, images can be suboptimal and usually requires an extra visit prior to implantation, therefore an intraprocedural way of identifying the optimal areas could be beneficial.

It is not known whether lead position as targeted by imaging methods of mechanical activation corresponds to the site of latest electrical activation, nor whether sensed electrical signals correspond to sites of scar. Investigators are planning to investigate the relationship between the site of latest mechanical activation using TTE and the site of latest electrical activation of the LV; and between scar and sensed electrical signals.

If the area of latest mechanical activation is related to the area of latest electrical activation then this can be an alternative, more convenient and cost effective way of assessing optimal LV lead positioning.

ELIGIBILITY:
Inclusion Criteria:

1. LV Ejection Fraction ≤ 35 %
2. New York Heart Association class I-IV
3. QRS ≥130ms
4. Left Bundle Branch Block
5. Male or female, aged 18 years or above
6. Able to give consent

Exclusion Criteria:

1. Patients with Atrial Fibrillation
2. Unable to give consent
3. QRS≤120 ms
4. Right Bundle Branch Block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HF, LBBB and have been referred for CRT.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Q-LV (electrical activation of the left ventricle) at different sites of the left ventricle | 1 day
  The time from onset of depolarisation (Q wave) to sensed electrogram in the left ventricle ("LV") will be measured at various sites over the left ventricular epicardium to build up a map of myocardial electrical activation

SECONDARY OUTCOMES:
Mechanical activation of the left ventricle using echocardiography | 1 day
  The pattern of mechanical activation of the left ventricle will be determined using speckle-tracking echocardiography.

IPD SHARING:
Plan to Share IPD: No